CLINICAL TRIAL: NCT07369661
Title: A Brief Self-compassion Intervention for Body Image, Minority Stress, and Sexual Self-efficacy in Hong Kong Gay Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HE-NHS2025/05; M2025/06 (Other Grant/Funding Number: Hong Kong Metropolitan University)
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gay Men
Keywords: gay men; self-compassion; body image; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We will include a self-compassion intervention group and a waiting-list control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion interventional group (Experimental): Interventional group will include 2.5 hour training and 3 weeks self-compassion writing exercise
  Interventions: Behavioral: Brief self-compassion intervention
- Waiting-list control group (No Intervention): Waiting-list control group

INTERVENTIONS:
Behavioral: Brief self-compassion intervention — Participants will be randomly allocated to the self-compassion group and the waiting list control group. The interveintion group will receive a 2.5 self-compassion training, and 3 week self-compassion writing exercise.
  Arms: Self-compassion interventional group

SUMMARY:
This pilot study aims to explore the feasibility, acceptability, and preliminary effectiveness of a brief self-compassion writing intervention on body image, minority stress, and sexual self-efficacy among gay men in Hong Kong.

DETAILED DESCRIPTION:
Gay men experience greater body dissatisfaction, a stronger drive for muscularity, and heightened body image concerns compared to their heterosexual counterparts. These issues contribute to minority stress, anxiety, low self-esteem, and engagement in risky sexual behaviors. Using a randomized controlled trial (RCT) design, we aim to explore the feasibility, acceptability, and preliminary effectiveness of a brief self-compassion writing intervention on body image, minority stress, and sexual self-efficacy among gay men in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* self-identified as a gay man
* sufficient comprehension of Cantonese
* currently living in Hong Kong
* able to provide informed consent

Exclusion Criteria:

* currently experiencing psychosis
* having an intellectual disability
* experiencing current suicidal ideation
* not currently receiving or engaging in regular mental health services in the last 3 months
* participation in a similar study or receiving similar services in the past 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study focuses on gay men.
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
self-compassion | From enrollment to the end of intervention at 1 month
  Self-compassion will be measured using the 12-item short version of the self-compassion scale (SCS). Items are rated on a 5-point Likert scale ranging from 1 (Almost Never) to 5 (Almost Always). The total score ranged from 12 to 60, with higher score indicating higher level of self-compassion.

SECONDARY OUTCOMES:
Sexuality-based stigma | From enrollment to the end of treatment at 1 month
  Sexuality-based stigma will be measured by the 10-item Chinese men sex with men (MSM) Stigma Scale. Items are rated on a four-point Likert scale from 1 (never) to 4 (many times). The total score ranges from 10 to 40, with higher score indicating higher level of sexuality-based stigma.
Internalized stigma | From enrollment to the end of treatment at 1 month
  Internalized stigma will be measured with the 5-item revised internalized homophobia scale (IHP-R). Items are measured on a five-point Likert scale between 1 (Strongly Disagree) and 5 (Strongly Agree). The total score ranges from 5 to 25, with higher scores indicate greater internalized stigma.
anxiety | From enrollment to the end of treatment at 1 month
  Anxiety symptoms will be measured using the 7-item Generalized Anxiety Disorder-7 (GAD-7). Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher total scores indicating higher levels of anxiety symptoms
self-esteem | From enrollment to the end of treatment at 1 month
  The 10-item Rosenberg Self-Esteem Scale (RSE) will be used to measured self-esteem. Items will be rated on a 4-point Liker scale (1 = Strongly agree, 4 = Strongly disagree). The total score ranges from 10 to 40, with higher score indicating higher level of self-esteem.
body objectification | From enrollment to the end of treatment at 1 month
  Self-objectification will be measured using the Chinese version of the Objectified Body Consciousness Scale (OBCS) - body-surveillance subscale. It consists of eight items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree). The total score ranges from 7 to 56, with a higher score indicating a higher level of body surveillance.
sexual self-efficacy | From enrollment to the end of treatment at 1 month
  The 14-item Condom Self-Efficacy Scale (CSES) will be used to measurement participants' sexual self-efficacy. Items will be measured on a 5-point Likert scale, ranging from 1 (very unsure) to 5 (very sure). The total score ranging from 14 to 70, with higher scores indicated a higher level of condom use efficacy.
Body shame | From enrollment to the end of intervention at 1 month
  Body shame will be measured using the Chinese version of the Objectified Body Consciousness Scale (OBCS) - body shame subscale (McKinley & Hyde, 1996). It consists of six items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with a higher score indicating a higher level of body shame.
Depression | From enrollment to the end of intervention at 1 month
  Depression will be measured using the Chinese version of the 9-item Patient Health Questionnaire (PHQ-9). Items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher total scores indicating higher levels of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided